CLINICAL TRIAL: NCT07059949
Title: Phase II, Single-center Study of Short-course Radiotherapy Followed by CAPOX and Carrelizumab and Bevacizumab or Cetuximab in the Treatment of Initially Unresectable Metastatic Rectal Cancer
Brief Title: Short Course Radiotherapy Followed by CAPOX and Carrilizumab and Bevacizumab or Cetuximab for the Initial Treatment of Unresectable Metastatic Rectal Cancer
Acronym: Union-mRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Union-mRC(ongoing)
Record Dates: First submitted 2025-04-17; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Unresectable Metastatic Rectal Cancer; CAPOX; Combination of Radioimmunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Can't remove RAS/BRAF completely wild (Experimental): CAPOX+ Camrelizumab + Cetuximab
  Interventions: Drug: CAPOX+ Camrelizumab+ Cetuximab
- RAS/BRAF mutations cannot be resected (Experimental): CAPOX+ Camrelizumab + Bevacizumab
  Interventions: Drug: CAPOX+ Camrelizumab+ Bevacizumab

INTERVENTIONS:
Drug: CAPOX+ Camrelizumab+ Cetuximab — For advanced primary treatment of unresectable rectal cancer, primary radiation therapy DT 25Gy/5F, and rest for 1 week, followed by CAPOX chemotherapy + Camrelizumab + Bevacizumab or Cetuximab (KRAS, NRAS, and BRAF all wild-type Cetuximab, KRAS, NRAS, and BRAF variants selected Bevacizumab) for 4-6 months, after which Capecitabine + Camrelizumab + Bevacizumab or Cetuximab was maintained
  Arms: Can't remove RAS/BRAF completely wild
Drug: CAPOX+ Camrelizumab+ Bevacizumab — For advanced primary treatment of unresectable rectal cancer, primary radiation therapy DT 25Gy/5F, and rest for 1 week, followed by CAPOX chemotherapy + Camrelizumab + Bevacizumab or Cetuximab (KRAS, NRAS, and BRAF all wild-type Cetuximab, KRAS, NRAS, and BRAF variants selected Bevacizumab) for 4-6 months, after which Capecitabine + Camrelizumab + Bevacizumab or Cetuximab was maintained
  Arms: RAS/BRAF mutations cannot be resected

SUMMARY:
To evaluate the efficacy and safety of short-course radiotherapy followed by CAPOX and carrilizumab and bevacizumab or cetuximab in the initial treatment of unresectable metastatic rectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent and be able to comply with the visiting arrangements and related procedures stipulated in the programme;
2. Age ≥18 years old and ≤75 years old, gender is not limited;
3. Histologically confirmed rectal cancer with initial treatment (no surgery, radiotherapy, chemotherapy, targeted therapy or immunotherapy);
4. Radiologically confirmed unresectable metastatic rectal cancer (cTxNxM1);
5. Tissue samples must be provided for molecular typing (such as PD-L1, MSI, KRAS, NRAS, BRAVF, etc.), and newly acquired groups are preferred For patients who cannot provide newly obtained tissue, 5-8 paraffin sections with a thickness of 5um can be provided for archiving.
6. No serious abnormality of blood system, heart, lung, liver, kidney function and immune deficiency;
7. Baseline * (within 7 days before the first administration of the study drug) blood routine tests meet the following requirements:

   Hemoglobin ≥90g/L Absolute neutrophil count (ANC) ≥1.5×109

   /L Platelet count ≥100×109/L Eosinophils ≤1.5× Upper limit of normal (ULN)

   * Throughout the protocol, "baseline" is defined as the last available observation before the first administration of the investigational drug. Subjects must not have received blood transfusion products (including red suspension, apheresis platelets, cryoprecipitate, etc.), erythropoietin, or colony-stimulating factor support therapy within 7 days prior to blood sample collection.
8. Serum biochemical tests at baseline (within 7 days before the first dose) met the following requirements

   Requirements:

   Total bilirubin ≤1.5× Upper limit of normal (ULN) (if total bilirubin > 1.5× upper limit of normal, combined with bilirubin

   ≤ULN was allowed to be included in the study); Aspartate aminotransferase (AST) or Alanine aminotransferase (AST) ALT) ≤2.5× upper limit of normal value; Serum Creatinine ≤1.5×ULN or Clearance of Creatinine (CCr) ≥45mL/min were obtained by Cockcroft-Gault formula Calculate CCr (using actual body weight); Albumin ≥30g/L.
9. Coagulation tests at baseline (within 7 days before the first dose) meet the following requirements:

   International normalizaed ratio (INR) ≤1.5×ULN (≤3× if receiving steady dose anticoagulation therapy) ULN); Partial thromboplastin time (PTT) (or activated partial plastin time (PTT)) thromboplastin time, aPTT]) ≤1.5×ULN (≤3×ULN if receiving stable dose anticoagulant therapy);
10. Urine routine examination at baseline (within 7 days before the first dose) meets the following requirements: urinary protein (UPRO) < 2+ or 24-hour urinary protein quantity < 1g;
11. At least one measurable lesion according to RECIST v1.1 (Solid tumor) criteria;
12. The Physical status score (ECOG PS) of the Eastern United States Tumor Consortium was 0 or 1;
13. Expected survival time ≥3 months.
14. Female subjects of childbearing age or male subjects whose partner is a female of childbearing age agree to strictly use effective contraception throughout the treatment period and for 6 months after the treatment period

Exclusion Criteria:

1. Previous exposure to any anti-PD-1 or anti-PD-L1 antibodies;
2. Women who are breastfeeding, pregnant or preparing to become pregnant;
3. Corticosteroid (dose equivalent to prednisone >10 mg/ day) or other immunosuppressive therapy should be administered within 2 weeks prior to study drug administration;
4. Active, known, or suspected autoimmune disease or previous 2-year history of the disease (vitiligo, psoriasis, alopecia, or Grave's disease that did not require systemic treatment within the last 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type 1 diabetes requiring only insulin replacement therapy were eligible);
5. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation; People with HIV, or active hepatitis B or C (active hepatitis B reference: ≥104 copies /ml of HBV DNA; Active hepatitis C reference: HCV RNA≥103 copies /ml);
6. Interstitial lung disease (including past and present disease), such as interstitial pneumonia, pulmonary fibrosis, or evidence of ILD on baseline chest CT or MRI;
7. Allergy and multiple drug allergy;
8. There are serious heart, lung, liver and kidney dysfunction, such as decompensated heart, lung, kidney, liver and other major organ dysfunction, failure or poor blood sugar control, can not tolerate chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to initial efficacy evaluation,assessed up to 6 months
  Objective response rate

SECONDARY OUTCOMES:
PFS | From enrollment to the first appearance of disease progression or date of deathfrom any cause,whichever came first, assessed up to 18 months
  Progression free survival
OS | From enrollment to patient death,assessed up to 36 months
  Overall Survival
DCR | Through out the study (24 months)
  Disease Control Rate
Adverse Event (AE), Treatment-Emergent AE (TEAE), Adverse Event of SpecialInterest (AESl) and Serious Adverse Event (SAE) | Through out the study (up to 36 months)
  Adverse events will be assessed by investigator(s) according to CommonTerminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).